CLINICAL TRIAL: NCT04834557
Title: Evaluating the Effect of Digoxin and Ursodeoxycholic Acid in Patients With Rheumatoid Arthritis in Egypt
Brief Title: Evaluating the Effect of Digoxin and Ursodeoxycholic Acid in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mariam George Tadros Bolous, Assistant Lecturer of Clinical pharmacy, Faculty of Pharmacy, Sinai University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Treating Rheumatoid Arthritis
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Digoxin; Ursodeoxycholic acid; Synovial inflammation; leukocyte infiltration; Autoimmune diseases; Th17 and Treg cells; Synovial hypoxia
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases | interventions — Digoxin; Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Participants in this arm will receive Placebo with the current DMARDs treatments for rheumatoid arthritis for 24 weeks.
  Interventions: Drug: Placebo
- Digoxin (Experimental): Participants in this arm will receive digoxin 0.25 mg every other day + DMARDs for 24 weeks.
  Interventions: Drug: Digoxin 0.25 mg
- Ursodeoxycholic acid (UDCA) (Experimental): Participants in this arm will receive ursodeoxycholic acid (UDCA) 500 mg/day + DMARDs for 24 weeks.
  Interventions: Drug: Ursodeoxycholic acid (UDCA) 500 mg

INTERVENTIONS:
Drug: Placebo — Placebo will be administered to the control group for 24 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Control
Drug: Digoxin 0.25 mg — All subjects will receive digoxin administered at 0.25 mg every other day for 24 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Digoxin
Drug: Ursodeoxycholic acid (UDCA) 500 mg — All subjects will receive Ursodeoxycholic acid (UDCA) administered at 500 mg/day for 24 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Ursodeoxycholic acid (UDCA)

SUMMARY:
The purpose of this study is to investigate the potential therapeutic effects of the cardiac glycoside digoxin and the secondary bile acid ursodeoxycholic acid (UDCA) on synovial inflammation and disease activity when administered as add-on treatments to the current DMARDs treatments for rheumatoid arthritis patients with variant disease activity.

DETAILED DESCRIPTION:
This study is a randomized, open-labeled, controlled prospective study to evaluate the potential therapeutic effects of the cardiac glycoside digoxin and the secondary bile acid ursodeoxycholic acid (UDCA) on synovial inflammation and disease activity when administered as add-on treatments to the current DMARDs treatments for rheumatoid arthritis patients with variant disease activity. The study population will be rheumatoid arthritis patients attending the Physical Medicine, Rheumatology and Rehabilitation Department at Menoufia University Hospital, Menoufia, Egypt. A total of 90 rheumatoid arthritis patients who will meet the inclusion criteria will be enrolled in this study. The 90 participants will be divided into 30 rheumatoid arthritis patients who will receive placebo + the current DMARDs treatments of rheumatoid arthritis for 24 weeks and serve as the control group, 30 rheumatoid arthritis patients who will receive DMARDs + digoxin 25 mg every other day for 24 weeks and the last 30 rheumatoid arthritis patients who will receive DMARDs + ursodeoxycholic acid (UDCA) 500 mg/day for 24 weeks. Clinical Examinations and laboratory parameters will be performed and measured at the beginning of the study, 12 weeks and 24 weeks after randomization to evaluate the efficacy of digoxin and UDCA in the treatment of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis according to the ACR/EULAR 2010 criteria.
* Having active rheumatoid arthritis disease activity (the 28-joint disease activity score [DAS28] according to the CRP formula > 2.6).
* Aged between 18 and 80 years.
* With clear consciousness and able to cooperate with this study.
* Personal willingness and ability to comply with the study follow-up schedule and other requirements of the study protocol.
* Both male and female will be included
* All patients receiving non-biological drugs will be also included.
* Sign an informed consent for the clinical study.

Exclusion Criteria:

* Pregnant or planning to be pregnant and breast-feeding women
* Patients suffering from any chronic diseases
* Patients with other autoimmune diseases, such as systemic lupus erythematosus, Sjogren's syndrome and mixed connective tissue disease.
* Patients who have a diagnosis of any other inflammatory arthritis (e.g., psoriatic arthritis or ankylosing spondylitis).
* Patients with a history of, or suspected, demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis).
* Patients with a current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
* Patients treated with biological therapy such as TNF-α or IL-1β antagonists.
* Patients with infectious or inflammatory diseases, endocrine disorders, any past or current psychiatric or neurological diseases.
* Patients with cardiovascular diseases such as arrhythmias and acute myocardial infarction.
* Patients with electrolyte disturbances (such as hypokalemia, hypomagnesemia, and hypercalcemia) could potentially elevate the risk of digoxin toxicity.
* Patients with clinically significant hepatic and renal dysfunction or impairment.
* Alcohol abuse
* Patients with evidence of viral (HBV or HCV), autoimmune hepatitis, and decompensated liver disease.
* Patients with cancer currently diagnosed or in medical history, if no recovery was achieved.
* Patients who are allergic to digoxin or Ursodeoxycholic acid (UDCA)
* Patients who are unconscious and unable to complete the study.
* Patients with acute inflammation of the gall bladder or the biliary tract, frequent episodes of biliary colic, and impaired contractility of the gall bladder, will be excluded.
* Patients with cholestasis, primary biliary cirrhosis, or biliary obstruction will also be excluded.
* Patients who have received an organ transplant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Clinical Disease Activity Index (CDAI) Score | Baseline, after 12 weeks, after 24 weeks
  To evaluate the effect of the use of digoxin and UDCA as an add-on therapy in patients with rheumatoid arthritis by evaluating the change from baseline in the clinical findings as measured by Clinical Disease Activity Index (CDAI) scores. A lower CDAI score from Baseline would mean improvement in disease activity and an increase in CDAI score from Baseline would mean an increase in disease activity or a worsening in disease activity. Scores: 0.0-2.8 = Range for Remission; 2.9-10.0 = Range for Low disease activity; 10.1-22.0 Range for Moderate disease activity; 22.1-76 Range for High disease activity. Total range is from 0-100, with the high scores representing high disease activity.
Changes in C-Reactive Protein (CRP) Values and Erythrocyte Sedimentation Rates (ESR) | Baseline, after 12 weeks, after 24 weeks
  C- reactive Protein (CRP) values and Erythrocyte Sedimentation Rate (ESR) will be made at baseline and after 12 as well as 24 weeks to determine the number of patients whose test result improved or worsened CRP value (normal range <1.0 mg/dl). ESR (normal range 0-28 mm/hr) . If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.

SECONDARY OUTCOMES:
Changes from baseline Measurement of IL-17A and HIF-1α at 12 and 24 weeks | Baseline, after 12 weeks, after 24 weeks
  Serum IL-17A and HIF-1α levels will be measured by means of the human enzyme-linked immunosorbent assay (ELISA) technique according to the manufacturer's protocol.
Numbers of participants with treatment-related adverse events | Baseline, after 12 weeks, after 24 weeks
  The adverse events in each group will be observed and documented during the whole procedure to show the safety of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nageh Ahmed El-Mahdy, Professor, Study Chair — Professor of Pharmacology and Toxicology Faculty of Pharmacy, Tanta University; Medhat Ismail Abdel Hamid, Professor, Study Chair — Professor of Pharmacology and Toxicology Faculty of Medicine, Al-Azhar University; Dalia Salah Seif, PHD, Study Director — Associate Professor of Physical Medicine, Rheumatology and Rehabilitation Faculty of Medicine, Menoufyia University; Enass Yousef Osman, PHD, Study Director — Lecturer of Pharmacology and toxicology, Faculty of Pharmacy, Tanta University; Mariam George Tadros Bolous, Master, Principal Investigator — Assistant Lecturer of Clinical pharmacy, Faculty of Pharmacy, Sinai University
Locations (1):
- Menoufia University Hospital, Shibīn al Kawm, Egypt

REFERENCES:
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Neogi T, Aletaha D, Silman AJ, Naden RL, Felson DT, Aggarwal R, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Khanna D, Kvien TK, Laing T, Liao K, Mease P, Menard HA, Moreland LW, Nair R, Pincus T, Ringold S, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G; American College of Rheumatology; European League Against Rheumatism. The 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for rheumatoid arthritis: Phase 2 methodological report. Arthritis Rheum. 2010 Sep;62(9):2582-91. doi: 10.1002/art.27580. PMID 20872596
- [Background] Hua S, Dias TH. Hypoxia-Inducible Factor (HIF) as a Target for Novel Therapies in Rheumatoid Arthritis. Front Pharmacol. 2016 Jun 27;7:184. doi: 10.3389/fphar.2016.00184. eCollection 2016. PMID 27445820
- [Background] Lee EJ, Kwon JE, Park MJ, Jung KA, Kim DS, Kim EK, Lee SH, Choi JY, Park SH, Cho ML. Ursodeoxycholic acid attenuates experimental autoimmune arthritis by targeting Th17 and inducing pAMPK and transcriptional corepressor SMILE. Immunol Lett. 2017 Aug;188:1-8. doi: 10.1016/j.imlet.2017.05.011. Epub 2017 May 21. PMID 28539269
- [Background] O'Dwyer AM, Lajczak NK, Keyes JA, Ward JB, Greene CM, Keely SJ. Ursodeoxycholic acid inhibits TNFalpha-induced IL-8 release from monocytes. Am J Physiol Gastrointest Liver Physiol. 2016 Aug 1;311(2):G334-41. doi: 10.1152/ajpgi.00406.2015. Epub 2016 Jun 23. PMID 27340129
- [Background] Saeed H, Mateen S, Moin S, Khan AQ, Owais M. Cardiac glycoside digoxin ameliorates pro-inflammatory cytokines in PBMCs of rheumatoid arthritis patients in vitro. Int Immunopharmacol. 2020 May;82:106331. doi: 10.1016/j.intimp.2020.106331. Epub 2020 Feb 24. PMID 32106058
- [Derived] El-Mahdy NA, Tadros MG, El-Masry TA, Binsaleh AY, Alsubaie N, Alrossies A, Abd Elhamid MI, Osman EY, Shalaby HM, Saif DS. Efficacy of the cardiac glycoside digoxin as an adjunct to csDMARDs in rheumatoid arthritis patients: a randomized, double-blind, placebo-controlled trial. Front Pharmacol. 2024 Oct 21;15:1445708. doi: 10.3389/fphar.2024.1445708. eCollection 2024. PMID 39498340